CLINICAL TRIAL: NCT06766838
Title: Outcomes Of The Different Techniques Of Male Circumcision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Bakr Ahmed, Resident of pediatric surgery at sohag university Hospitals, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Soh-Med--24-12-02MS
Record Dates: First submitted 2024-12-29; First posted 2025-01-09 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Prepuce; Accessory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1. Group A: Conventional dissection technique; (Active Comparator): In this group, circumcision is performed by the dorsal slit technique. A slit is made dorsally to the level of about 5 mm from the coronal sulcus, and the redundant foreskin and mucosa were excised circumferentially. Hemostasis is secured with ligation , and the cut edges are sutured
  Interventions: Procedure: 1. Conventional dissection technique (group A) :
- 2. Group B: Bone cutting ; (Active Comparator): Two mosquito forceps are used to grasp the foreskin. The glans penis is squeezed back to avoid its injury. After that, bone cutting forceps is applied to the foreskin for 3 minutes, at the level of the mark, then the foreskin is excised by scalpel at the same level. Bleeding points are ligated and the cut edges are sutured with absorbable suture
  Interventions: Procedure: 2. Bone cutting forceps technique (Group B)
- 3. Group C: Electro-cauterization (bipolar) assisted circumcision; (Active Comparator): The skin is held by two hemostats to elevate the foreskin, and then the kocher clamp applied at the level of the skin to be removed for circumcision. Excess foreskin will be cut by scissor with hemostasis by bipolar cauterization.
  Interventions: Procedure: 3. Electro-cauterization (bipolar) assisted circumcision (Group C)
- 4. Group D: Thermal cauterization assisted circumcision; (Active Comparator): The skin is held by two hemostats to elevate the foreskin, and then the kocher clamp applied at the level of the skin to be removed for circumcision. Excess foreskin will be cut by thermal cauterization.
  Interventions: Procedure: 4. Thermal cauterization assisted circumcision (Group D)
- 5. Group E: Gomco clamp technique; (Active Comparator): The prepuce is grasped using two hemostats applied at 2 and 10 o'clock. A dorsal slit at 12 o'clock is made, and then the bell is applied gently to the glans. The base plate is placed over the metal bell. The foreskin then is protracted back over the bell with the clamps still attached. The foreskin is drawn evenly through the hole bilaterally using the ink mark as a guide. The clamp then is tightened and left in place for 5 minutes to squeeze the prepuce between the bell and the clamp to make it blood free before a circumferential incision is made.
  Interventions: Procedure: 5. Gomco clamp technique (Group E):
- 6. Group F: Plastibell device technique. (Active Comparator): The prepuce is grasped using two hemostats applied at 2 and 10 o'clock. A dorsal slit at 12 o'clock is made, appropriate-sized bell is placed over the glans, and the foreskin is brought over its top. The string is placed around the foreskin and the Plastibell device at the level of the mark in a groove that acted as the string placement guide. The string is then tightened and tied in a simple square knot. The excess foreskin is trimmed from around the bell using iris scissors.
  Interventions: Procedure: 6. Plastibell device technique (Group F):

INTERVENTIONS:
Procedure: 1. Conventional dissection technique (group A) : — In this group, circumcision is performed by the dorsal slit technique. A slit is made dorsally to the level of about 5 mm from the coronal sulcus, and the redundant foreskin and mucosa were excised circumferentially. Hemostasis is secured with ligation , and the cut edges are sutured with absorbable suture. Then, dressing is applied.
  Arms: 1. Group A: Conventional dissection technique;
Procedure: 2. Bone cutting forceps technique (Group B) — Two mosquito forceps are used to grasp the foreskin. The glans penis is squeezed back to avoid its injury. After that, bone cutting forceps is applied to the foreskin for 3 minutes, at the level of the mark, then the foreskin is excised by scalpel at the same level. Bleeding points are ligated and the cut edges are sutured with absorbable suture. Then, a dressing is applied
  Arms: 2. Group B: Bone cutting ;
Procedure: 3. Electro-cauterization (bipolar) assisted circumcision (Group C) — The skin is held by two hemostats to elevate the foreskin, and then the kocher clamp applied at the level of the skin to be removed for circumcision. Excess foreskin will be cut by scissor with hemostasis by bipolar cauterization.
  The skin retracted proximally after that to expose the glans. Sutures are made if there is separation between the skin and the mucous membrane.
  Arms: 3. Group C: Electro-cauterization (bipolar) assisted circumcision;
Procedure: 4. Thermal cauterization assisted circumcision (Group D) — The skin is held by two hemostats to elevate the foreskin, and then the kocher clamp applied at the level of the skin to be removed for circumcision. Excess foreskin will be cut by thermal cauterization. The skin retracted proximally after that to expose the glans. Sutures are made if there is separation between the skin and the mucous membrane.
  Arms: 4. Group D: Thermal cauterization assisted circumcision;
Procedure: 5. Gomco clamp technique (Group E): — The prepuce is grasped using two hemostats applied at 2 and 10 o'clock. A dorsal slit at 12 o'clock is made, appropriate-sized bell is placed over the glans, and the foreskin is brought over its top. The string is placed around the foreskin and the Plastibell device at the level of the mark in a groove that acted as the string placement guide. The string is then tightened and tied in a simple square knot. The excess foreskin is trimmed from around the bell using iris scissors. The handle is then broken off the device
  Arms: 5. Group E: Gomco clamp technique;
Procedure: 6. Plastibell device technique (Group F): — The prepuce is grasped using two hemostats applied at 2 and 10 o'clock. A dorsal slit at 12 o'clock is made, appropriate-sized bell is placed over the glans, and the foreskin is brought over its top. The string is placed around the foreskin and the Plastibell device at the level of the mark in a groove that acted as the string placement guide. The string is then tightened and tied in a simple square knot. The excess foreskin is trimmed from around the bell using iris scissors. The handle is then broken off the device
  Arms: 6. Group F: Plastibell device technique.

SUMMARY:
Aim of work:

The aim of study is to comprehensively evaluate and compare the efficacy, safety, clinical outcomes, cosmetic appearance and complication rates associated with different technique of circumcisions.

DETAILED DESCRIPTION:
The aim of study is to comprehensively evaluate and compare the efficacy, safety, clinical outcomes, cosmetic appearance and complication rates associated with different technique of circumcisions.

Patients and methods:

According to the method of circumcision used; infants were divided into 5 groups :

1. Group A: Conventional dissection technique;
2. Group B: Bone cutting ;
3. Group C: Electro-cauterization (bipolar) assisted circumcision;
4. Group D: Thermal cauterization assisted circumcision;
5. Group E: Gomco clamp technique;
6. Group F: Plastibell device technique. Place of the study: The study will be held in the department of Pediatric surgery at Sohag University Hospital.

Type of the study: Prospective comparative Cohort study. Duration of the study: The study lasts for 6 months from the acceptance of the protocol (december 2024) to (Jone 2025).

Inclusion criteria:

All uncircumcised boys with intact prepuce aged below 15 years presented at our department for routine circumcision or for medical indications.

Exclusion criteria:

1. Age above 15 years
2. Ambiguous genitalia
3. Congenital penile anomalies e.g. hypospadias, epispadias, buried penis, webbed penis, micropenis, congenital chordee, incomplete prepuce and mega-urethra.
4. Redo-circumcision
5. Balanitis or inflammatory process around the penis.
6. Bleeding disorders; hemophilia or thrombocytopenia

ELIGIBILITY:
Inclusion Criteria:

1. All uncircumcised boys with intact prepuce
2. Age below 5 years presented at our department for routine circumcision or for medical indications.

Exclusion Criteria:

1. Age above 5 years
2. Ambiguous genitalia
3. Congenital penile anomalies
4. Redo-circumcision
5. Balanitis or inflammatory process around the penis.
6. Bleeding disorders

Max Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Bleeding | 1 day
  combine the number of dressing, Significant bleeding is considered if the dressing is completely soaked

SECONDARY OUTCOMES:
Cosmetic appearance | 1 month
  Score for parent and physician
  * Excellent 3
  * Good 2
  * Poor 1

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] [1] Myers A, Earp B. What Is the Best Age to Circumcise? A Medical and Ethical Analysis. Bioethics. 2020;34:645-663. [2] Schneider, T., 2013. Ancient Egypt investigated: 101 important questions and intriguing answers. Bloomsbury Publishing. [3] Alanis MC, Lucidi RS. Neonatal circumcision: a review of the world's oldest and most controversial operation. Obstet Gynecol Surv 2004;59(5):379e95. [4] Abdulwahab-Ahmed, A. and Mungadi, I.A., 2013. Techniques of male circumcision. Journal of surgical technique and case report, 5(1), pp.1-7. [5] Deacon, M. and Muir, G., 2023. What is the medical evidence on non-therapeutic child circumcision?. International journal of impotence research, 35(3), pp.256-263. [6] Iacob, S.I., Feinn, R.S. and Sardi, L., 2022. Systematic review of complications arising from male circumcision. BJUI compass, 3(2), pp.99-123. [7] Prakash, K.P., 2019. Comparative Study of Frenulum Sparing Circumcision with Dorsal Slit-Sleeve Technique of Circumcision for Phimosis (Master's thesis, Rajiv Gandhi University of Health Sciences (India). [8] Prabhakaran S, Ljuhar D, Coleman R, Nataraja RM. Circumcision in the paediatric patient: a review of indications, technique and complications. J Paediatr Child Health. 2018;54(12):1299-307. [9] Zafar, G.M., Sajjad, M.N., Zaheer, M., Yousaf, M.H. and Javeed, M.N., 2024. Split Glans & Advancement Flap To Repair Penile Hair Tourniquet Injury In Children: A Challenging Problem Of Unknown Etiology. Pakistan Journal of Urology (PJU), 2(01), pp.82-87. [10] Wang X, Dong C, Beekoo D et al. (2019): Dorsal penile nerve block via perineal approach, an alternative to a caudal block for pediatric circumcision: a randomized controlled trial. BioMed Research International, 19:6875756. doi: 10.1155/2019/6875756. [11] Kamil M (2012): Bone cutter circumcision in neonates. AL-Kindy College Medical Journal, 8(1): 119-121. [12] Wan J (2002): Gomco circumcision clamp: an enduring and unexpected success. Urology, 59(5): 790- 794. [13] Morris B, Eley C (2011): Male circumcision: An appraisal of current instrumentation. Biomedical Engineering, University of Rijeka, Rijeka, Pp. 315-354. DOI: 10.5772/18543